CLINICAL TRIAL: NCT01835327
Title: Cerebral Oximetry and Recovery Following Thoracic Surgery
Brief Title: Cerebral Oxygen Monitoring During Surgery and Recovery After Surgery in Patients Having Lung Surgery
Status: Terminated | Type: Observational
Why Stopped: PI no longer at institution
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Other Study IDs: GCO 12-1398; HS#: 12-00716
Record Dates: First submitted 2013-04-16; First posted 2013-04-18 (Estimated); Last update posted 2017-02-15 (Actual); Status verified 2017-02

CONDITIONS: Cerebral Oxygen Desaturation
Keywords: intraoperative, post-operative recovery; thoracic surgery; cerebral oximetry

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Exposed: Cerebral oximetry desaturation below 65% for a minimum of 3 minutes
- Not Exposed: Those patients who do not experience a cerebral oxygen desaturation below 65% for a minimum of 3 minutes

SUMMARY:
The current study proposes to address the question of whether patients' cerebral oxygen saturation levels are predictive of their recovery from thoracic surgery. Further, the study poses the hypothesis that a patient's poor recovery status goes on to increase a patient's risk of developing post-operative morbidities such as pneumonia, arrhythmias and delirium. The aim of this study is to address the observation that some patients struggle more than others in their recovery and that 1) this may be a result of intraoperative cerebral oxygen desaturations and 2) that this may affect their post-operative morbidity. If a potential means of predicting poor outcomes is identified this will lead to further research into how to adjust the associated variables, such as cerebral oxygenation, to improve patient post-operative outcome.

DETAILED DESCRIPTION:
Despite advances in the field of thoracic surgery, post-operative morbidity continues to be a significant problem with limited understanding of the connection between the insult of surgery and anesthesia and the pathophysiology of the development of these morbidities. Surgeons in the thoracic department have noted that some patients seem to recover less vigorously than other patients. What accounts for these different recovery trajectories is unclear. Researchers have developed a Post-Operative Quality Recovery Scale (PQRS) which assesses six domains (physiologic, nociceptive, emotive, activities of daily living, cognitive, and overall patient experience) and has been suggested to serve as a means of tracking patients' recovery from surgery.

ELIGIBILITY:
Inclusion Criteria:

* speak English
* 18 yo or older
* willing to participate
* undergoing thoracic surgery at Mount Sinai Hospital that will require one lung ventilation

Exclusion Criteria:

* prisoners
* lack capacity to consent to trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Anticipated inclusion is all patients scheduled for thoracic surgery at Mount Sinai Hospital by the aforementioned surgeons Dr. Flores and Dr. Kaufman. Exclusion criteria will be those patients who (1) do not speak English, (2) are less that the age of 18 years old, (3) are currently prisoners, (4) do not display the capacity to consent to the trial and (5) who are unwilling to complete the study. Screening for exclusion criteria will occur primarily in the pre-operative setting under the guidance of Drs. Flores and Kaufman and will be reviewed by the Research Coordinator and acting anesthesiologist on the day of surgery.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Post-Operative Quality of Recovery Score (PQRS) | up to 3 months
  Patients are assessed 30 minutes, one hour, and three hours post extubation time on day of surgery and then once daily for however long they are hospitalized up to 14 days, patients are then assessed via phone at one month and three months post-op. Recovery is assessed via questions on multiple domains such as pain and nausea, emotional status, activities of daily living and cognitive status.
Post-Operative Morbidity Survey (POMS) Score | Post-Operative day 3
  The POMS score measures morbidity across multiple categories with pre-defined thresholds, example: Pulmonary (de novo requirement of oxygen supplementation), Infectious (fever above 38C or require antibiotics) etc.
Post-Operative Morbidity Survey (POMS) Score | Post-Operative day 5
  The POMS score measures morbidity across multiple categories with pre-defined thresholds, example: Pulmonary (de novo requirement of oxygen supplementation), Infectious (fever above 38C or require antibiotics) etc.
Post-Operative Morbidity Survey (POMS) Score | Post-Operative day 8
  The POMS score measures morbidity across multiple categories with pre-defined thresholds, example: Pulmonary (de novo requirement of oxygen supplementation), Infectious (fever above 38C or require antibiotics) etc.

SECONDARY OUTCOMES:
Cognitive Assessment Method | up to 14 days
  Also measuring delirium each day of hospitalization POD1-POD14 via modified and validated version of the CAM (Cognitive Assessment Method).

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Silverstein, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Monique Roberts, BA, Study Director — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

REFERENCES:
- [Background] Royse CF, Newman S, Chung F, Stygall J, McKay RE, Boldt J, Servin FS, Hurtado I, Hannallah R, Yu B, Wilkinson DJ. Development and feasibility of a scale to assess postoperative recovery: the post-operative quality recovery scale. Anesthesiology. 2010 Oct;113(4):892-905. doi: 10.1097/ALN.0b013e3181d960a9. PMID 20601860
- [Background] Daubeney PE, Pilkington SN, Janke E, Charlton GA, Smith DC, Webber SA. Cerebral oxygenation measured by near-infrared spectroscopy: comparison with jugular bulb oximetry. Ann Thorac Surg. 1996 Mar;61(3):930-4. doi: 10.1016/0003-4975(95)01186-2. PMID 8619720
- [Background] Goldman S, Sutter F, Ferdinand F, Trace C. Optimizing intraoperative cerebral oxygen delivery using noninvasive cerebral oximetry decreases the incidence of stroke for cardiac surgical patients. Heart Surg Forum. 2004;7(5):E376-81. doi: 10.1532/HSF98.20041062. PMID 15799908
- [Background] Murkin JM, Adams SJ, Novick RJ, Quantz M, Bainbridge D, Iglesias I, Cleland A, Schaefer B, Irwin B, Fox S. Monitoring brain oxygen saturation during coronary bypass surgery: a randomized, prospective study. Anesth Analg. 2007 Jan;104(1):51-8. doi: 10.1213/01.ane.0000246814.29362.f4. PMID 17179242
- [Background] Slater JP, Guarino T, Stack J, Vinod K, Bustami RT, Brown JM 3rd, Rodriguez AL, Magovern CJ, Zaubler T, Freundlich K, Parr GV. Cerebral oxygen desaturation predicts cognitive decline and longer hospital stay after cardiac surgery. Ann Thorac Surg. 2009 Jan;87(1):36-44; discussion 44-5. doi: 10.1016/j.athoracsur.2008.08.070. PMID 19101265
- [Background] Hemmerling TM, Bluteau MC, Kazan R, Bracco D. Significant decrease of cerebral oxygen saturation during single-lung ventilation measured using absolute oximetry. Br J Anaesth. 2008 Dec;101(6):870-5. doi: 10.1093/bja/aen275. Epub 2008 Oct 3. PMID 18835887
- [Background] Bennett-Guerrero E, Welsby I, Dunn TJ, Young LR, Wahl TA, Diers TL, Phillips-Bute BG, Newman MF, Mythen MG. The use of a postoperative morbidity survey to evaluate patients with prolonged hospitalization after routine, moderate-risk, elective surgery. Anesth Analg. 1999 Aug;89(2):514-9. doi: 10.1097/00000539-199908000-00050. PMID 10439777
- [Background] Grocott MP, Browne JP, Van der Meulen J, Matejowsky C, Mutch M, Hamilton MA, Levett DZ, Emberton M, Haddad FS, Mythen MG. The Postoperative Morbidity Survey was validated and used to describe morbidity after major surgery. J Clin Epidemiol. 2007 Sep;60(9):919-28. doi: 10.1016/j.jclinepi.2006.12.003. Epub 2007 May 7. PMID 17689808
- [Background] Ackland GL, Harris S, Ziabari Y, Grocott M, Mythen M; SOuRCe Investigators. Revised cardiac risk index and postoperative morbidity after elective orthopaedic surgery: a prospective cohort study. Br J Anaesth. 2010 Dec;105(6):744-52. doi: 10.1093/bja/aeq245. Epub 2010 Sep 28. PMID 20876700
- [Background] Ackland GL, Moran N, Cone S, Grocott MP, Mythen MG. Chronic kidney disease and postoperative morbidity after elective orthopedic surgery. Anesth Analg. 2011 Jun;112(6):1375-81. doi: 10.1213/ANE.0b013e3181ee8456. Epub 2010 Aug 31. PMID 20807976
- [Background] Hollowell J, Grocott MP, Hardy R, Haddad FS, Mythen MG, Raine R. Major elective joint replacement surgery: socioeconomic variations in surgical risk, postoperative morbidity and length of stay. J Eval Clin Pract. 2010 Jun;16(3):529-38. doi: 10.1111/j.1365-2753.2009.01154.x. Epub 2010 Feb 18. PMID 20210822
- [Background] Davies SJ, Yates D, Wilson RJ. Dopexamine has no additional benefit in high-risk patients receiving goal-directed fluid therapy undergoing major abdominal surgery. Anesth Analg. 2011 Jan;112(1):130-8. doi: 10.1213/ANE.0b013e3181fcea71. Epub 2010 Nov 3. PMID 21048092
- [Background] Grichnik KP, Ijsselmuiden AJ, D'Amico TA, Harpole DH Jr, White WD, Blumenthal JA, Newman MF. Cognitive decline after major noncardiac operations: a preliminary prospective study. Ann Thorac Surg. 1999 Nov;68(5):1786-91. doi: 10.1016/s0003-4975(99)00992-3. PMID 10585059
- [Background] Murkin JM. Cerebral oximetry: monitoring the brain as the index organ. Anesthesiology. 2011 Jan;114(1):12-3. doi: 10.1097/ALN.0b013e3181fef5d2. No abstract available. PMID 21178667
- [Background] Tang L, Kazan R, Taddei R, Zaouter C, Cyr S, Hemmerling TM. Reduced cerebral oxygen saturation during thoracic surgery predicts early postoperative cognitive dysfunction. Br J Anaesth. 2012 Apr;108(4):623-9. doi: 10.1093/bja/aer501. Epub 2012 Feb 5. PMID 22311364
- [Background] Kazan R, Bracco D, Hemmerling TM. Reduced cerebral oxygen saturation measured by absolute cerebral oximetry during thoracic surgery correlates with postoperative complications. Br J Anaesth. 2009 Dec;103(6):811-6. doi: 10.1093/bja/aep309. PMID 19918024
- [Background] Sauer AM, Kalkman C, van Dijk D. Postoperative cognitive decline. J Anesth. 2009;23(2):256-9. doi: 10.1007/s00540-009-0744-5. Epub 2009 May 15. PMID 19444566
- [Background] Fischer GW, Benni PB, Lin HM, Satyapriya A, Afonso A, Di Luozzo G, Griepp RB, Reich DL. Mathematical model for describing cerebral oxygen desaturation in patients undergoing deep hypothermic circulatory arrest. Br J Anaesth. 2010 Jan;104(1):59-66. doi: 10.1093/bja/aep335. PMID 19933513
- [Background] Fischer GW, Torrillo TM, Weiner MM, Rosenblatt MA. The use of cerebral oximetry as a monitor of the adequacy of cerebral perfusion in a patient undergoing shoulder surgery in the beach chair position. Pain Pract. 2009 Jul-Aug;9(4):304-7. doi: 10.1111/j.1533-2500.2009.00282.x. Epub 2009 Mar 17. PMID 19490464
- [Background] Fischer GW, Stone ME. Cerebral air embolism recognized by cerebral oximetry. Semin Cardiothorac Vasc Anesth. 2009 Mar;13(1):56-9. doi: 10.1177/1089253208330710. Epub 2009 Jan 27. PMID 19174527
- [Background] Fischer GW, Lin HM, Krol M, Galati MF, Di Luozzo G, Griepp RB, Reich DL. Noninvasive cerebral oxygenation may predict outcome in patients undergoing aortic arch surgery. J Thorac Cardiovasc Surg. 2011 Mar;141(3):815-21. doi: 10.1016/j.jtcvs.2010.05.017. Epub 2010 Jun 25. PMID 20579669